CLINICAL TRIAL: NCT06880783
Title: Effect of Manual Diaphragmatic Release Technique on Exercise Capacity and Sleep Quality in Older Adults With Type II Diabetes: a Randomized Controlled Trial
Brief Title: Manual Diaphragmatic Release Technique on Exercise Capacity and Sleep Quality
Acronym: DM and sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, Lecturer of Physical therapy, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Diabetes and Sleep Quality
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Active Comparator): Participants will receive manual diaphragm release technique combined with deep breathing exercises
  Interventions: Other: manual diaphragm release technique; Other: deep breathing exercises
- Control group (Active Comparator): Participants will receive deep breathing exercises
  Interventions: Other: deep breathing exercises

INTERVENTIONS:
Other: manual diaphragm release technique — The participant should be supine with relaxed limbs, and the therapist should position themselves at the head, making manual contact with the pisiform, hypothenar region, and fingers. The therapist should gently pull the contact towards the head, deepen it during exhalation, and gradually increase the depth.
  Arms: Study Group
Other: deep breathing exercises — Participants in a crook laying position are instructed to inhale through the nose, lift the abdomen, and let out through the mouth, breathing six breaths per minute for 30 minutes.

SUMMARY:
To investigate if there is a significant effect of manual diaphragmatic release technique on exercise capacity, sleep quality, chest expansion, ADL, fatigue and quality of life in older adults with type II diabetes.

DETAILED DESCRIPTION:
Participants, including both genders, will have a history of Diabetes Type II for more than one year. They will be well controlled with HbA1c≤7. Patients will be aged from 55 years and above and had a body mass index less than 30 kg/m². Patients will follow up on the training program and instructions. They will be medically stable.

ELIGIBILITY:
Inclusion Criteria:

* History of Diabetes Type II for more than one year.
* They will be well controlled with HbA1c≤7.
* Patients will be aged from 55 years and above and had a body mass index less than 30 kg/m².
* Patients will follow up on the training program and instructions. They will be medically stable.

Exclusion Criteria:

* Chest diseases.
* Diaphragmatic hernia, clinical evidence of phrenic nerve injury, recent abdominal or thoracic surgery, or history of traumatic lesion possibly affecting diaphragm.
* History of Myocardial infarction and/or cardiothoracic surgery
* Unstable medical status.
* Cognitive disability hindering responding to the questionnaires.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | up to 6 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Pittsburgh Sleep Quality Index (PSQI) | up to 6 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete

CONTACTS AND LOCATIONS:
Locations (1):
- Beni suef hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No